CLINICAL TRIAL: NCT01661218
Title: Complications and Risk Factors Related With Central Venous Catheters in Cancer Patients(CVCCP)
Brief Title: Complications and Risk Factors Related With Central Venous Catheters in Cancer Patients
Acronym: CVCCP
Status: Completed | Type: Observational
Sponsor: Beijing Huanxing Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCH20120530; HCH20120530-008 (Other: Beijing Huanxing Cancer Hospital)
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2012-08

CONDITIONS: Thrombosis; Infections
Keywords: catheters; Central Venous; complications; cancer
MeSH Terms: conditions — Thrombosis; Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- complications: catheter-related venous thrombosis catheter-related infections

SUMMARY:
The investigators aim to determine the complications and risk factors related with peripherally inserted central catheters (PICCs) and central venous catheters (CVCs) in cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine the complications and risk factors related with peripherally inserted central catheters (PICCs) and central venous catheters (CVCs) in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* all adult cancer patients with central venous catheters (CVCs) or peripherally inserted central catheters (PICCs) placed at BeijingHCH.

Exclusion Criteria:

* without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult cancer patients with CVC and PICC placed at BeijingHCH and with written consent for this study
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2012-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Catheter-related venous thrombosis and catheter-related infections | 30 days after PICC and CVC line withdrawn
  Catheter-related venous thrombosis and catheter-related infections

SECONDARY OUTCOMES:
Catheter tip position | participants will be followed before PICC and CVC line withdrawn
  Catheter tip position

CONTACTS AND LOCATIONS:
Overall Officials: Jian DING, MD, Study Chair — Beijing Huanxing Cancer Hospital
Locations (1):
- Beijing Huanxing Cancer Hospital, Beijing, Beijing Municipality, China